CLINICAL TRIAL: NCT06244602
Title: Balance Assessment in Individuals With Chronic Pain: an Explorative Study of Psychometric Properties of the Mini-BESTest
Brief Title: Test-retest and Experiences During Balance Assessment With the Mini-BESTest
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Pernilla Asenlof, Professor, Uppsala University
Other Study IDs: 2023-04206-01
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Non-Cancer Pain
Keywords: Postural Balance; Chronic pain; Psychometrics; Experiences; Test-retest
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test psychometric properties of a clinical balance assessment scale, the Mini-BESTest, as well as to explore experiences and beliefs about balance and being balance tested. The main research questions are:

* What is the test-retest reliability of the Mini-BESTest balance assessment scale for individuals with long-term pain?
* What is the individual's subjective beliefs and experiences about their own balance and being balance tested with the Mini-BESTest?

Tow samples of participants will be included. One sample for a) the test-retest evaluation or b) an interview during and after performing the Mini-BESTest.

DETAILED DESCRIPTION:
Individuals with chronic pain, i.e., pain > 3 months, report balance problems and falls in their everyday lives. How balance affects daily functioning, and how to identify individuals with balance impairments are less studied. The Mini-BESTest has previously shown adequate construct validity in individuals with chronic pain, however, the test-retest reliability has not been explored. There is also a need of studies that have focus on the person's own experiences of balance and the balance tested.

In this observational study we aim to examine the psychometric properties of the Mini-BESTest, in individuals with chronic pain. Further we aim to explore individual subjective beliefs and experiences about own balance and being balance tested.

A convenience selection will be used to include two samples of participants. One sample for the test-retest evaluation, here after called the test-retest part of the study. And one sample for a think aloud interview, here after called the interview part of the study. At baseline the participants will be included to one of the two parts.

Participants in the test-retest part will be assessed with the Mini-BESTest on two occasions, the baseline and the re-test within approximately 2 weeks. The inclusion to the test-retest sample will continue until at least 50 individuals with no subjective experience of improvement or deterioration in balance status between the first and second occasions, according to the self-report measure the Patient global impression of change (PGIC), are included. This sampling is done in purpose to calculate test-retest reliability in individuals without subjective change in balance between the two occasions.

To the interview part, approximately ten to twenty individuals will be included for concurrent think aloud, i.e., think aloud during balance testing with the Mini-BESTest, and recurrent think aloud, i.e., an interview after the balance assessment. The interviews will cover questions about the participants experience of the testing with the Mini-BESTest and their balance.

Data will be collected by use of digitized questionnaires, physical performance tests, a structured interview and data from medical records.

Statistical tests will be used to evaluate test-retest reliability and internal consistency. The interviews will be analyzed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* pain duration of 3 months or more
* a visit for investigation or treatment at the pain clinic

Exclusion Criteria:

* receiving acute care related to active cancer treatment
* receiving palliative care
* having cognitive impairments
* illiterate in the Swedish language
* wheelchair users or bed-bound
* current participating in any of the rehabilitation programs at the pain clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include individuals with chronic pain referred to or in specialized pain care.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
The Mini Balance Evaluation Systems Test (Mini-BESTest) | Baseline, 2 weeks
  Self-report, Swedish version. Dynamic balance is measured with 14 items ranging from 0 = 'unable or requiring help to perform' to 2 = 'normal'. All items are summed up to a total score which ranges from 0 to 28, with higher scores reflecting better balance.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | Baseline, 2 weeks
  Self-report, oral question. Current pain intensity is measured with a scale that ranges from 0-10, where 0 = 'no pain' and 10 = 'pain as bad as can be'.
Fall frequency | Baseline, 2 weeks
  Self-report, question about fall frequencies over the last previous year and the last three weeks.
Activities-Specific Balance Confidence (ABC) scale | Baseline, 2 weeks
  Self-report, Swedish version. Balance confidence is measured with 16 items ranging from 0 = 'No confidence' to 100 = 'Full confidence'. All items are summed up to a total score, which ranges from 0 to 100, with higher scores reflecting higher balance confidence while doing activities.
Falls Efficacy Scale - international (FES-I) | Baseline, 2 weeks
  Self-report, Swedish version. Fear of falling is measured with 16 items ranging from 1 = 'Not at all concerned' to 4 = 'Very concerned'. All items are summed up to a total score, which ranges from 16 to 64, with higher scores reflecting more concerns about falling.
Numerical Rating Scales (NRS) | Baseline
  Self-report. Pain severity is measured with four scales where worst, least, average and current pain during the past week are scored. Each scale ranges from 0-10, where 0 = 'no pain' and 10 = 'pain as bad as can be'.
The Pain Disability Index (PDI) | Baseline
  Self-report, Swedish version. Pain-related disability is measured with 7 items measuring family/home responsibilities, recreation, social activity, occupation, sexual behavior, self-care and life support activity. Every item ranges from 0 = 'No disability' to 10 = 'Worst disability'. All seven items are summed up in a total score, which ranges from 0 to 70, with higher scores reflecting higher interference of pain with daily activities.
2-item Pain Self-Efficacy Questionnaire (PSEQ-2) | Baseline
  Self-report, Swedish version. Pain self-efficacy is measured with 2 items ranging from 0 = 'Not at all confident' to 6 = ' Completely confident', with a higher combined scores indicating stronger self-efficacy beliefs.
11-item Tampa Scale for Kinesiophobia (TSK-11) | Baseline
  Self-report, Swedish version. Fear of movement and reinjury is measured by 11 items ranging from 1 = 'Does not agree at al' to 4 = 'totally agree). A total score is calculated ranging from 11 to 44 where higher scores indicates higher fear of movement.
The Public Health Agency of Sweden' questions about physical activity | Baseline
  Self-report. Minutes of physical activity on low intensity and moderate intensity is measured with two ordinal scales.
Question about sedentary from the Swedish National Board of Health and Welfare | Baseline
  Self-report. Hours of sedentary behavior measured on an ordinal scale.
The Time Line Follow-Back (TLFB) Structured interview | Baseline
  Patterns of opioid use (type of opioid, dose, and duration) will be measured using a structured interview, calendar format, using 4 weeks intervals starting with the most recent complete week, week 1, working backward one week at time recording days of use for each opioid.

OTHER OUTCOMES:
Patient global impression of change (PGIC) | 2 weeks
  Self-report. The measure reflects participant's beliefs about if there balance has changed between baseline and the re-test of Mini-BESTest. The participant indicates whether he/she feels that his/her balance has changed since the previous session of the study on a 7-point scale, 'very much improved', 'much improved', 'minimally improved', 'no change', 'minimally worse', 'much worse', 'very much worse'.
Change in medication | 2 weeks
  Self-report questions on change in medication between baseline and the re-test of the Mini-BESTest. The participant indicates whether the type of medication or dose has changed since the previous study visit, the name of the changes medicine, and whether the medicine has been 'added' or 'removed', as well as if the dose has 'increased', 'decreased' or if the participant 'doesn't know'.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Professor, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Uppsala University and University Hospital, Uppsala, Sweden